CLINICAL TRIAL: NCT03667508
Title: Evaluation the Efficacy of Rapid and Slow Maxillary Expansion in Posterior Crossbite Treatment Using Cone Beam Computed Tomography
Brief Title: Effectiveness of Rapid and Slow Maxillary Expansion in Treating Posterior Crossbite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-19-2018
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Posterior Crossbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid Maxillary Expansion (Experimental): Patients will undergo Rapid Maxillary Expansion using a rapid maxillary expanding device, i.e. a Hyrax expander (modified by McNamra).
  Interventions: Procedure: Rapid Maxillary Expanding Device
- Slow Maxillary Expansion (Active Comparator): Patients will undergo Slow Maxillary Expansion using a slow maxillary expanding device, i.e. a removable appliance with a central screw.
  Interventions: Procedure: Slow Maxillary Expanding Device

INTERVENTIONS:
Procedure: Rapid Maxillary Expanding Device — The expansion screw will be turned two times in the first day, and then daily until the correction is achieved.
  Other Names: Bonded Acrylic Hyrax Expander
  Arms: Rapid Maxillary Expansion
Procedure: Slow Maxillary Expanding Device — The expansion screw will be activated every five days until correcting the crossbite.
  Other Names: Removable Expansion Plate
  Arms: Slow Maxillary Expansion

SUMMARY:
This study will evaluate the efficacy of rapid maxillary expansion (RME) and slow maxillary expansion (SME) in treating posterior crossbite using cone beam computed tomography.

The study sample will consist of 32 patients who suffer from a skeletal posterior crossbite. The sample will be allocated randomly into two groups: RME group and SME group.

The skeletal and dento-alveolar changes occurring after treatment will be assessed by using cone beam computed tomography(CBCT) radiographs.

DETAILED DESCRIPTION:
Unilateral or bilateral posterior crossbite (PXB) is a common malocclusion. In recent decades, RME has gained preference as the treatment of choice for PXB. However, the side effects, such as reported pain, relapse of the expansion, tipping of the molars, bone loss, gingival recession, and root resorption, have lead some clinicians to prefer SME.

In this study the investigators will treat PXB using two techniques, RME and SME. Patients will be divided into two groups (a technique in each group) to evaluate the efficacy of each one using cone beam computed tomography.

RME group: A Hyrax appliance modified as McNamara will be applied. SME group: A removable appliance with central expander will be applied. In order to evaluate the changes occurring, two CBCT radiography will be taken for every individual: first, before treatment, second, after three months of retention for RME group and one month of retention for SME group

ELIGIBILITY:
Inclusion Criteria:

* Bilateral skeletal maxillary deficiency (symmetrical) which will be clinically and radiographically diagnosed.
* Bilateral or unilateral functional posterior crossbite ( combined with mandibular shifting)
* Class I or II malocclusion.
* Normal or slight vertical growth pattern.

Exclusion Criteria:

* Poor oral hygiene.
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Patients with low facial height.
* A contraindication for rapid or slow maxillary expansion procedures.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-06-15 (Actual)

PRIMARY OUTCOMES:
Change in the mandibular path of closure | T0: one day before the commencement of treatment; T1: after the end of active treatment and a retention period (which is expected within 14-15 weeks in the rapid expansion group and within 16-20 weeks in the slow expansion group)
  The path of the lower jaw from the rest position until closure will be clinically examined.
  The path is classified as
  1. normal path of closure
  2. deviated path of closure due to premature contacts
Change in the anterior maxillary expansion width | T0: one day before the commencement of treatment; T1: after the end of active treatment and a retention period (which is expected within 14-15 weeks in the rapid expansion group and within 16-20 weeks in the slow expansion group)
  This will be assessed using cone-beam computed tomography. The anterior maxillary expansion width is measured between RPyP-LPyP (RPyP: Right piriform point. The most lateral and caudal point of the nasal piriform aperture, at the boundary with the palatal cortex. LPyP: Analogue to RPyP, left side)
Change in the posterior expansion width | T0: one day before the commencement of treatment; T1: after the end of active treatment and a retention period (which is expected within 14-15 weeks in the rapid expansion group and within 16-20 weeks in the slow expansion group)
  This will be assessed using cone-beam computed tomography. The posterior maxillary expansion width is measured between RPaFoP and LPaFoP (RPaFoP: Right palatine foramen point. The most posterior point of the right greater palatine foramen in the maxilla within the palatal cortex. LPaFoP: Analogue to RPaFOPr, left side.)
Change in the Pterygoid expansion width | T0: one day before the commencement of treatment; T1: after the end of active treatment and a retention period (which is expected within 14-15 weeks in the rapid expansion group and within 16-20 weeks in the slow expansion group)
  This will be assessed using cone-beam computed tomography. The Pterygoid expansion width is measured between PtR and PtL on the images. (PtR. Pterygoideous right. The most caudal point of the apex of the right pterygoid process of the sphenoid. PtL. Pterygoideous left. Analogue to PtR, left side)
Change in the inter-molar width | T0: one day before the commencement of treatment; T1: after the end of active treatment and a retention period (which is expected within 14-15 weeks in the rapid expansion group and within 16-20 weeks in the slow expansion group)
  This will be assessed using cone-beam computed tomography. The inter-molar width is measured at molar cusps between the right and left teeth.
Change in molar tipping | T0: one day before the commencement of treatment; T1: after the end of active treatment and a retention period (which is expected within 14-15 weeks in the rapid expansion group and within 16-20 weeks in the slow expansion group)
  This will be measured in cone-beam computed tomography images. Molar tipping is defined as the difference between (AR-AL) and (CR-CL) CR:Cuspid right which is the mesio-palatal cusp tip of the right maxillary first molar, whereas CL: Cuspid left which is the mesiopalatal cusp tip of the left maxillary first molar.
  AR: Apex right which is the apex of the palatal root of the right maxillary first molar, where as AL: Apex left which is the apex of the palatal root of the left maxillary first molar.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Rabah, DDS, Principal Investigator — MSc student at the Orthodontic Department, University of Damascus Dental School, Damascus, Syria; Mohammad Y Hajeer, DDS MSc PhD, Study Director — Associate Professor of Orthodontics, University of Damascus Dental School, Damascus, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martina R, Cioffi I, Farella M, Leone P, Manzo P, Matarese G, Portelli M, Nucera R, Cordasco G. Transverse changes determined by rapid and slow maxillary expansion--a low-dose CT-based randomized controlled trial. Orthod Craniofac Res. 2012 Aug;15(3):159-68. doi: 10.1111/j.1601-6343.2012.01543.x. Epub 2012 Mar 27. PMID 22812438
- [Background] Greenbaum KR, Zachrisson BU. The effect of palatal expansion therapy on the periodontal supporting tissues. Am J Orthod. 1982 Jan;81(1):12-21. doi: 10.1016/0002-9416(82)90283-4. PMID 6758588
- [Background] Sandikcioglu M, Hazar S. Skeletal and dental changes after maxillary expansion in the mixed dentition. Am J Orthod Dentofacial Orthop. 1997 Mar;111(3):321-7. doi: 10.1016/s0889-5406(97)70191-4. PMID 9082855
- [Background] Brunetto M, Andriani Jda S, Ribeiro GL, Locks A, Correa M, Correa LR. Three-dimensional assessment of buccal alveolar bone after rapid and slow maxillary expansion: a clinical trial study. Am J Orthod Dentofacial Orthop. 2013 May;143(5):633-44. doi: 10.1016/j.ajodo.2012.12.008. PMID 23631965
- [Background] Bucci R, D'Anto V, Rongo R, Valletta R, Martina R, Michelotti A. Dental and skeletal effects of palatal expansion techniques: a systematic review of the current evidence from systematic reviews and meta-analyses. J Oral Rehabil. 2016 Jul;43(7):543-64. doi: 10.1111/joor.12393. Epub 2016 Mar 23. PMID 27004835
- [Derived] Rabah N, Al-Ibrahim HM, Hajeer MY, Ajaj MA. Evaluation of rapid versus slow maxillary expansion in early adolescent patients with skeletal maxillary constriction using cone-beam computed tomography: A short-term follow-up randomized controlled trial. Dent Med Probl. 2022 Oct-Dec;59(4):583-591. doi: 10.17219/dmp/133513. PMID 36108265